CLINICAL TRIAL: NCT04296266
Title: Human Salivary Gland Disposition of Alda-341 in Patients Undergoing Salivary Gland Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-32994
Record Dates: First submitted 2020-02-20; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-02

CONDITIONS: Submandibular Gland Tumor; Parotid Gland Tumor
MeSH Terms: conditions — Submandibular Gland Neoplasms; Parotid Neoplasms | interventions — Limonene

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Alda-341 treatment (Experimental): Alda-341 treatment at 2 g/day for 14 days up until the day before regular medical care surgery.
  Interventions: Drug: Alda-341

INTERVENTIONS:
Drug: Alda-341 — Dietary supplement d-limonene orally administered as a drug.
  Other Names: d-limonene

SUMMARY:
The purpose of this study is determine salivary gland disposition of d-limonene, the primary component in citrus peel and a common dietary supplement.

Salivary gland tissue and saliva will be collected to determine concentration of d-limonene and its metabolites in these tissues.

DETAILED DESCRIPTION:
Primary Objective: To determine the bioavailability of Alda-341 in salivary gland tissue.

Secondary Objective: To determine the bioavailability of Alda-341 in saliva and blood

ELIGIBILITY:
Inclusion Criteria:

* Elected to undergo surgery for recent diagnosis of parotid or submandibular gland tumor
* Ability to adhere to study visit schedule and other protocol requirements
* Operable candidate base on the surgeon's note
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Nursing or pregnant
* Diagnosis of kidney disease, history of renal disease with creatinine > 1.5 mg/dL, or currently on dialysis
* Diagnosis of end stage liver disease
* Any unstable medical condition
* Use of chemotherapy or radiotherapy within 4 weeks before first dose of study dietary supplement
* Unwilling to stop dietary supplements 3 weeks before first dose of study dietary supplement

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Bioavailability of Alda-341 in salivary gland tissue using GCMS | 2 week
  Bio availability of Alda-341 in salivary gland tissue will be measured using gas chromatography mass spectrometry (GCMS). The scale is is 4ng/mL - 8000ng/mL.

SECONDARY OUTCOMES:
Bioavailability of Alda-341 in saliva and blood | 2 week
  Bio availability of Alda-341 in saliva and blood will be measured using gas chromatography mass spectrometry (GCMS). The scale is is 4ng/mL - 8000ng/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Quynh-Thu Le, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No